CLINICAL TRIAL: NCT05992740
Title: The Optimal Sequence of Bronchial Brushing, Forceps Biopsy and Washing for Diagnosis of Lung Cancer
Brief Title: Role of Bronchoscope in Diagnosis of Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Maged Monir, principal investigator, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: bronchoscope in lung cancer
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopes

STUDY DESIGN:
Intervention Model Description: analytical cross sectional
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bronchial wash group (Active Comparator): the patients will undergo bronchoscope then pre-biopsy bronchial wash, biopsy, post-biopsy bronchial wash will be obtained
  Interventions: Device: bronchoscope
- bronchial brush (Active Comparator): the patients will undergo bronchoscope then pre-biopsy bronchial brush, biopsy, post-biopsy bronchial brush will be obtained
  Interventions: Device: bronchoscope

INTERVENTIONS:
Device: bronchoscope — bronchoscpe with broncial brush and biopsy or bronchial wash and biopsy

SUMMARY:
The study aims to compare the diagnostic yields of bronchial brushing performed before and after forceps biopsy and bronchial wash performed before and after biopsy during flexible bronchoscopy.

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer-related mortality in both sexes in the world. To treat the disease successfully, it should be diagnosed at the earliest possible stage. Several studies have demonstrated that early detection, localization, and aggressive treatment of lung cancer result in the 5-year survival rate of 70-80%. Nowadays, bronchoscopy is an invaluable tool for diagnosis of lung cancer and various diagnostic tools have been developed using flexible fiber-optic bronchoscopy (FOB).

Bronchoscopy, while essential for diagnosing and staging lung cancer, can give variable diagnostic yields ranging from37-77%. One reason for this variability is limitations in tissue sampling techniques, which can make it impossible to obtain the most representative area of neoplastic tissue. Numerous basic diagnostic procedures using FB, including bronchoalveolar lavage or washing, brushing, endobronchial or transbronchial biopsy(TBB), and transbronchial needle aspiration, have been evaluated in various combinations to improve the diagnostic yield of FB in patients with suspected lung cancer. However, the optimum sequence of brushing, washing and biopsy samples for diagnosing peripheral lung cancer is not clear and requires further study.

ELIGIBILITY:
Inclusion Criteria:

Patients in whom clinical findings, radiological examination suggested lung malignancy. patients with chronic cough, hemoptysis and lymph node enlargement.

Exclusion Criteria:

patients with no evidence of malignancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
comparison between diagnostic yields of different tissue sampling techniques of bronchoscope in lung cancer diagnosis | 2 years
  we will compare between the diagnostic yield of bronchial brushing group (pre-biopsy brushing + forceps biopsy + post-biopsy brushing) with the diagnostic yield of bronchial wash group (pre-biopsy bronchial wash + biopsy + post-biopsy bronchial wash).

REFERENCES:
- [Background] Hou G, Miao Y, Hu XJ, Wang W, Wang QY, Wu GP, Wang EH, Kang J. The optimal sequence for bronchial brushing and forceps biopsy in lung cancer diagnosis: a random control study. J Thorac Dis. 2016 Mar;8(3):520-6. doi: 10.21037/jtd.2016.02.12. PMID 27076949
- [Background] Lim JH, Kim MJ, Jeon SH, Park MH, Kim WY, Lee M, Kim JH, Kim JS, Kim YS, Kim L, Lee KH, Kwak SM, Shin H, Nam HS. The optimal sequence of bronchial brushing and washing for diagnosing peripheral lung cancer using non-guided flexible bronchoscopy. Sci Rep. 2020 Jan 23;10(1):1036. doi: 10.1038/s41598-020-58010-w. PMID 31974454